CLINICAL TRIAL: NCT05912452
Title: Investigation of the Effects of Vibration, Dynamic Stretching, and Kinesiotaping Applications on Proprioception, Muscle Strength, and Functional Parameters
Brief Title: Effects of Vibration, Stretching, and Taping on Proprioception, Strength, and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: bmenek...
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Stretch; Vibration; Disorder
Keywords: Vibration; Dynamic stretching; kinesiotape
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Percussion Massage Group (Experimental): The group to which percussion massage therapy will be applied to the deltoid muscle.
  Interventions: Other: Percussion Massage Therapy
- Kinesiotape Group (Experimental): The group to which kinesiotaping will be applied to the deltoid muscle.
  Interventions: Other: Kinesiotaping
- Dynamic Stretching Group (Experimental): The group to which dynamic stretching will be applied to the deltoid muscle.
  Interventions: Other: Dynamic stretching

INTERVENTIONS:
Other: Percussion Massage Therapy — Individuals who receive percussion massage therapy will be treated with a 5-minute medium-frequency percussion massage on the deltoid muscle group every other day. Percussion massage therapy will be applied in a total of 10 sessions and will be completed in 20 days.
  Arms: Percussion Massage Group
Other: Kinesiotaping — the Kinesiotape group; Kinesiotape banding will be done with 25% tension by applying a Y band to the deltoid muscle group. After the application, the Kinesio band will stay on the participant for 2 days. The next day, the participant will rest. This cycle will be repeated for 20 days.
  Arms: Kinesiotape Group
Other: Dynamic stretching — Dynamic stretching exercises will be applied to the shoulder flexor and abductor muscle groups in the Dynamic Stretching Group with 10 repetitions. As in percussion massage therapy, these exercises will be performed under the supervision of a physiotherapist every other day. The application will continue for 20 days.
  Arms: Dynamic Stretching Group

SUMMARY:
Percussion massage devices used in percussion massage therapy provide great convenience for both self-application and application by a physiotherapist.Percussion massage therapy is widely used today in many areas in deep and superficial tissues; such as pain reduction, increased blood circulation, improved scar tissue, reduced lactate levels and muscle spasms, increased lymphatic flow, inhibition of Golgi reflex, increased range of motion. There are deficiencies in the literature when studies related to these recently introduced devices are examined. To our knowledge, no study has been conducted so far that examines the immediate and short-term muscle strength, joint position sense, and functional parameters of percussion massage therapy.

Stretching exercises are used by athletes to increase joint range of motion and performance in the long term. It is also included in athletes' training programs for the purpose of warming up before an activity or cooling down after an activity. In many studies where the dynamic stretching method is affected, there are studies showing that dynamic stretching exercises performed before activity or sports positively affect performance and flexibility parameters. Therefore, many clinicians recommend dynamic stretching exercises before sports.Dr. Kase, who developed the kinesiology tape, says that taping the muscle is more effective compared to immobilizing the joint with tape. The elastic properties of the muscle are impaired by trauma and overuse.The possible mechanisms of action depend on the degree of tension used in taping can be listed as reducing inflammation and swelling by increasing circulation and creating cooling in the area by increasing the subcutaneous interstitial space with a lifting effect on the skin, increasing the signals sent to the central nervous system by stimulating the skin's mechanoreceptors and as a result, reducing pain with the gate control mechanism. When the literature is examined, it has been reported that Kinesiotape applications are not superior to other treatment modalities, but can be used to support treatment.Based on all this information, it is planned to investigate the immediate and short-term effects of percussion massage therapy, stretching exercises, and Kinesiotape applications in the literature."

DETAILED DESCRIPTION:
A total of 45 healthy individuals who meet the inclusion criteria will be included in the study at Istanbul Medipol University South Campus, Floor B4, Physiotherapy Practice Hall. Inclusion Criteria:

1. Those who can perform performance tests
2. Those who have not undergone orthopedic surgery from any region
3. Those without movement restriction
4. Individuals without a professional sports history will be included in the study.

Exclusion Criteria:

1. History of trauma
2. Anatomical deformities and skeletal system fractures
3. Diagnosed orthopedic or rheumatological diseases
4. Having been included in a physiotherapy program in the last 6 months
5. Individuals with pain in any region will be excluded from the study. Volunteer consent forms will be signed by individuals willing to participate in the study, and their demographic information will be recorded. 45 people will be included in the study and they will be divided into 3 groups.

1. Percussion Massage Therapy Group 2. Dynamic Stretching Group 3. Kinesiotape Group Individuals who receive percussion massage therapy will be treated with a 5-minute medium-frequency percussion massage on the deltoid muscle group every other day. Percussion massage therapy will be applied in a total of 10 sessions and will be completed in 20 days. - Dynamic stretching exercises will be applied to the shoulder flexor and abductor muscle groups in the Dynamic Stretching Group with 10 repetitions. As in percussion massage therapy, these exercises will be performed under the supervision of a physiotherapist every other day. The application will continue for 20 days. For the Kinesiotape group; Kinesiotape banding will be done with 25% tension by applying a Y band to the deltoid muscle group. After the application, the Kinesio band will stay on the participant for 2 days. The next day, the participant will rest. This cycle will be repeated for 20 days. Applications will be applied to the dominant shoulder of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Those who can perform performance tests
2. Those who have not undergone orthopedic surgery from any region
3. Those without movement restriction
4. Individuals without a professional sports history will be included in the study.

Exclusion Criteria:

1. History of trauma
2. Anatomical deformities and skeletal system fractures
3. Diagnosed orthopedic or rheumatological diseases
4. Having been included in a physiotherapy program in the last 6 months
5. Individuals with pain in any region will be excluded from the study.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Joint position sense | 10 minutes
  joint position sense will be evaluated with Becure Extremity ROM. Becure Extremity ROM is a technological system that allows for the objective measurement of joint range of motion by sensing reference points during extremity movements with its built-in camera and sensors. In the Becure Extremity ROM system, the patient is expected to stand in front of the camera and perform the desired movement. In the study, the ranges of motion for flexion and abduction of the shoulder joint will be recorded in degrees with Becure Extremity ROM. In the joint position sense measurements of the individuals participating in the study; individuals will first be asked to lift their shoulder to a certain degree, then bring it back to the same angle value while their eyes are closed. Joint position sense will be evaluated in terms of flexion and abduction. Differences in angle when eyes are closed and open will be recorded as joint position sense.
TFAST | 15 minutes
  Although there are arm and shoulder tests evaluating functional performance for athletes, performance tests commonly used to evaluate upper extremity functionality in a sedentary population or elderly individuals are not widespread. While joint range of motion (ROM) and strength evaluations are included in the tests used to assess upper extremity disorders, tests evaluating functional performance are often lacking. Or, many of the tests that include performance parameters target more functional individuals and ask them to take challenging starting positions, such as squat-jump or push-up. These tests are also not suitable for the majority of older populations with shoulder insufficiency, often along with other chronic musculoskeletal conditions. TFAST is a functional evaluation test that includes parameters such as joint range of motion, muscle strength, and endurance, and is particularly used for individuals who are not athletes.
Muscle Strenght | 5 minutes
  A dynamometer will be used to objectively measure the Deltoid muscle strength of all participants. The dynamometer is an assessment method that provides more sensitive results than manual muscle testing in objectively evaluating muscle strength. During the muscle strength measurement, the patient is first positioned. The dynamometer is then placed on the distal part of the area to be measured. The patient, on whom the force is applied, is asked to maintain their position. When the patient can no longer continue the movement, the application of force is stopped, and the maximum force recorded by the device is noted. Each measurement will be repeated three times, and the average of the test will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Merve YILMAZ MENEK, PhD, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No